CLINICAL TRIAL: NCT06755333
Title: Oral Hygiene Management of Hematologic Patients Undergoing Auto-transplantation: Observational Study
Brief Title: Oral Hygiene Management of Hematologic Patients Undergoing Auto-transplantation
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Rossana Izzetti, Researcher at the Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine of the University of Pisa, Principal Investigator, University of Pisa
Other Study IDs: 150782024
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic Stem Cell Transplantation; Dental Prophylaxis; Oral Hygiene; Motivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Oral hygiene motivation — the patient underwent a professional oral hygiene session before starting chemotherapy, as part of the routine pre-transplant procedure. Patients then received oral hygiene instructions.

SUMMARY:
This study assessed the effectiveness of a preventive protocol that included oral hygiene measures, patient education, and motivational strategies in individuals eligible for hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
At baseline (T0), the patient underwent a professional oral hygiene session prior to initiating chemotherapy, as part of the routine pre-transplant protocol. During this session, periodontal charting was completed, and patients were provided with oral hygiene instructions.

Following admission, patients received pre-transplant conditioning chemotherapy. Once engraftment of the transplant was confirmed by the Hematology Unit (9 days after engraftment), clinical parameters were reassessed (T1).

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* aged 18-75 years
* patients scheduled for HSCT
* acceptance of study participation
* compliance to follow-up

Exclusion Criteria:

- denial of the consent to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing autologous hematopoietic stem cell transplantation (HSCT) for hematologic diseases. The study included patients treated at the Hematology Unit of Pisa University Hospital. Participants were selected based on their eligibility for HSCT and their consent to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
PPD | measured at enrolment (T0) and 9 days after engraftment (T1)
  probing pocket depth (PPD) was measured as the distance from the free gingival margin to the bottom of the pocket by inserting a periodontal probe parallel to the longitudinal axis of the tooth using a periodontal probe (UNC 15, Hu-Friedy, Chicago, IL, USA) and a calibrated pressure of 0.3 N. All measurements were rounded to the nearest millimetre.
FMBS | measured at enrolment (T0) and 9 days after engraftment (T1)
  Full Mouth Bleeding Score (FMBS) was measured dichotomously after periodontal probing. The mean bleeding score was indicated as percentage of sites detected positive for bleeding on the total number of sites
FMPS | measured at enrolment (T0) and 9 days after engraftment (T1)
  Full Mouth Plaque Score (FMPS) was assessed the presence or absence of plaque on each tooth surface. The presence of plaque was evaluated as 1, while the absence as 0, on 6 sites per tooth (distobuccal, buccal, mesiobuccal, distolingual, lingual, mesiolingual). Mean plaque score was indicated as percentage of sites found positive for the presence of plaque on the total number of sites
CI | measured at enrolment (T0) and 9 days after engraftment (T1)
  Calculus Index was measured using a probe and considering supragingival and subgingival calculus separately, with score 0 assigned in the absence of calculus and score 3 assigned to supragingival calculus exceeding two-thirds of the crown and/or continuous bands of subgingival calculus
PRESENCE OF MUCOSITIS | measured 9 days after engraftment (T1)
  Presence of mucositis was evaluated as the presence of mucosal erythema or ulceration for 8 oral sites and assigning a score from 0 (normal oral mucosa) to 5 (>3 sites of ulceration).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine, University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No